CLINICAL TRIAL: NCT05038618
Title: A Phase II, Prospective, Open-Label, Single-Center Study to Evaluate the Safety, Tolerability, and Immunogenicity of COVID-19 Vaccine Candidate MVC-COV1901, CT-COV-21 Sub-study
Brief Title: A Study o Evaluate the Safety, Tolerability, and Immunogenicity of MVC-COV1901, CT-COV-21 Sub-study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT-COV-21s
Record Dates: First submitted 2021-08-25; First posted 2021-09-09 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2021-10

CONDITIONS: Covid19 Vaccine
Keywords: Covid19 vaccine
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MVC-COV1901(S protein with adjuvant) (Experimental): S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901(S protein with adjuvant)

INTERVENTIONS:
Biological: MVC-COV1901(S protein with adjuvant) — Approximately 400 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Day 1 and Day 29 via intramuscular (IM) injection in the deltoid region

SUMMARY:
This sub-study is a prospective open-label, single-center study to demonstrate comparability of different manufacturing scales.

DETAILED DESCRIPTION:
In this sub-study, approximately 400 adults participants who are generally healthy or with stable pre-existing health conditions aged ≥ 20 to < 65 years will be enrolled. The first 250 participants enrolled in this sub-study will receive MVC-COV1901(Scale A) and the remains will receive MVC-COV1901(Scale B). Each participant will receive 2 doses of study intervention, administered 28 days apart via IM injection in the deltoid region, preferably of the nondominant arm, at Day 1 and Day 29. The study procedure and visit schedule refer to the main study protocol and will be the same as the study procedure for the Immunogenicity Subset.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant ≥ 20 to < 65 years, or ≥ 65 years of age at randomization.
2. Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before enrollment and expected to remain stable for the duration of the study.
3. Female participant must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the last injection of study intervention. Acceptable forms include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c. Have a negative pregnancy test
4. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
5. Participant has not travelled overseas within 14 days of screening and will not have any oversea travelling throughout the study period.
6. Participant or the participant's legal representative must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding or have plan to become pregnant in 30 days after last administration of study intervention.
2. Employees at the investigator's site, of the Sponsor or the contract research organization (CRO) directly involved in the conduct of the study.
3. Currently receiving or received any investigational intervention within 30 days prior to the first dose of study intervention.
4. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the first dose of study intervention.
5. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the first dose of study intervention.
6. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of study intervention.
7. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the first dose of study intervention Medical Conditions
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarthritis, thyroiditis, Guillain-Barré syndrome, etc.).
11. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
12. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
13. Human immunodeficiency virus (HIV) antibody positive participants with CD4 count < 350 cells/mm3 or a detectable HIV viral load within the past year (low level variations from 50-500 viral copies/mL or equivalent which do not lead to changes in antiretroviral therapy [ART] are permitted).
14. Hepatitis B surface antigen (HBsAg) positive participant with positive hepatitis B e antigen (HBeAg) or abnormal liver function.
15. Hepatitis C virus (HCV) antibody positive participants with detectable HCV ribonucleic acid (RNA) viremia in recent 12 weeks.
16. Participant with ongoing acute diseases or serious medical conditions which will interfere with adherence to study requirements, or the evaluation of any study endpoint. Acute diseases or serious medical conditions include cardiovascular (e.g. New York Heart Association Grade III or IV), pulmonary (e.g. chronic obstructive pulmonary disease stage III or IV), hepatic (e.g. Child-Pugh Class C), neurologic (e.g. dementia), metabolic (e.g. diabetes mellitus with hemoglobin A1c [HbA1c] > 8%), renal (Stage 3 or worse chronic kidney disease), psychiatric condition (e.g. alcoholism, drug abuse), current severe infections, medical history, physical findings, or laboratory abnormality that in the investigators' opinion are not in stable condition and participating in the study could adversely affect the safety of the participant.

    Medigen Vaccine Biologics Corp. 34
17. Participant with previous known or potential exposure to SARS-CoV-1 or 2 viruses (EXCEPT for those who have been tested negative and completed the 14-day self-managements/ home quarantines/ home isolations) or received any other COVID-19 vaccine.
18. Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901.
19. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 399 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Event within 28 days post the second study intervention (Safety of MVC-COV1901) | Day 1 to 28 days after second vaccination
  To evaluate the safety and tolerability of MVC-COV1901 from Day 1 to 28 days after the second dose of study intervention in terms of the number and percentage of participants with the occurrence of:
  * Solicited local AEs (up to 7 days after each dose of study intervention)
  * Solicited systemic AEs (up to 7 days after each dose of study intervention)
  * Unsolicited AEs (up to 28 days after each dose of study intervention)
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901 | Day 1 to 28 days after second vaccination
  To evaluate the immunogenicity of MVC-COV1901among different manufacturing scales in terms of neutralizing antibody titers 28 days after the second vaccination

SECONDARY OUTCOMES:
Incidence of Adverse Event throughout study conduct (Safety of MVC-COV1901) | Day 1 to 180 days after second vaccination
  To evaluate the safety of MVC-COV1901 over the study period in terms of the number and percentage of participants with the occurrence of:
  * >= Grade 3 AE
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901 | Day 1 to 180 days after second vaccination
  To evaluate the immunogenicity of MVC-COV1901 among different manufacturing scales in terms of antigen-specific immunoglobulin and neutralizing antibody titers 28 days after the first dose of study intervention, 14 days after the second dose of study intervention, 28 days after the second dose of study intervention and 180 days after the second dose of study intervention

OTHER OUTCOMES:
Incidence of confirmed COVID-19 cases (Efficacy of MVC-COV1901) | Day 1 to 180 days after second vaccination
  To estimate the efficacy of MVC-COV1901, as compared to placebo, in the prevention of COVID-19 in terms of :
  * The number of laboratory-confirmed COVID-19 cases occurring ≥ 15 days after any dose of study intervention.
  * The number of laboratory-confirmed COVID-19 severe cases occurring ≥ 15 days after any dose of study intervention.
Cell-mediated immune response of MVC-COV1901 | Day 1 to 14 days after second vaccination
  To assess cell-mediated immune response of MVC-COV1901 as measured by intracellular cytokine staining (ICS) 28 days after the first dose of study intervention and 14 days after the second dose of study intervention
  -The percentage of specific cytokine response

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD, Principal Investigator — National Taiwan University Hospital; Tzou-Yien Lin, MD, Principal Investigator — Chang Gang Memorial Hospital, LinKou
Locations (1):
- Chang-Guang Memorial Hospital Lin-Kou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No